CLINICAL TRIAL: NCT03795584
Title: Endoclip Papillaplasty Restores Sphincter of Oddi Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Huang Yonghui, chief physician, Peking University Third Hospital
Other Study IDs: HYH20180520
Record Dates: First submitted 2018-06-12; First posted 2019-01-08 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Sphincter of Oddi Function

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoclip papillaplasty: Endoclip papilloplasty was performed to repair the Oddi sphincter using sterile repositionable hemostasis clipping device (Micro-tech (Nanjing), Co., Ltd.; stainless-steel). The participants underwent SOM before, immediately after EST, and 3 weeks after EST with endoclip papilloplasty. The participants were followed for 3 days during hospitalized.
  Interventions: Procedure: sterile repositionable hemostasis clipping device close the large duodenal papilla incision

INTERVENTIONS:
Procedure: sterile repositionable hemostasis clipping device close the large duodenal papilla incision — After the bile duct stent was placed, the investigators can use sterile repositionable hemostasis clipping device to close large duodenal papilla incision at 11 o'clock on the duodenal papilla.

SUMMARY:
Gallstones in the common bile duct (CBD) may be asymptomatic but may lead to complications such as acute cholangitis or acute pancreatitis. EST is widely used for the treatment of bile duct gallstones. Despite its efficacy and improvements over time, EST is still associated with complications such as hemorrhage, perforation, pancreatitis, and permanent loss of function of the sphincter of Oddi (SO). Permanent loss of SO function can cause duodenobiliary reflux, bacterial colonization of the biliary tract, gallstone recurrence, cholangitis, and liver abscess.

Endoscopic papillary balloon dilation (EPBD) was first proposed in 1983 and it is now recognized as an alternative technique for the removal of CBD gallstones. The small balloon (diameter <8 mm) is less invasive, reduces the occurrence of adverse effects, and preserves the SO function, but it has limitations in the presence of CBD gallstones ≥10 mm in diameter. EST combined with endoscopic papillary large-balloon dilation (EPLBD) has been introduced for patients with large gallstone, but EPLBD widens the distal common bile duct and still may cause SO function damage, partially or completely. Repairing the ampulla of Vater and SO may reduce the long-term complication rates, especially gallstone recurrence. Unfortunately, no efficient strategy has been proposed. The present pilot study aimed to examine the feasibility and efficiency of an innovative strategy named endoclip papilloplasty to repair the damaged ampulla and recover SO function. The advantage of this device is that it can be rotated clockwise or counterclockwise by turning the handle until the correct position is achieved. Another advantage is if the clip is not in desired position, it may be re-opened and repositioned. Once satisfying clip positioning is achieved, the clip can be firmly attached to the tissue by pulling the slider back until tactile resistance is felt in the handle.

DETAILED DESCRIPTION:
Gallstones in the common bile duct (CBD) may be asymptomatic but may lead to complications such as acute cholangitis or acute pancreatitis. EST is widely used for the treatment of bile duct gallstones. Despite its efficacy and improvements over time, EST is still associated with complications such as hemorrhage, perforation, pancreatitis, and permanent loss of function of the sphincter of Oddi (SO). Permanent loss of SO function can cause duodenobiliary reflux, bacterial colonization of the biliary tract, gallstone recurrence, cholangitis, and liver abscess.

Endoscopic papillary balloon dilation (EPBD) was first proposed in 1983 and it is now recognized as an alternative technique for the removal of CBD gallstones. The small balloon (diameter <8 mm) is less invasive, reduces the occurrence of adverse effects, and preserves the SO function, but it has limitations in the presence of CBD gallstones ≥10 mm in diameter. EST combined with endoscopic papillary large-balloon dilation (EPLBD) has been introduced for patients with large gallstone, but EPLBD widens the distal common bile duct and still may cause SO function damage, partially or completely. Repairing the ampulla of Vater and SO may reduce the long-term complication rates, especially gallstone recurrence. Unfortunately, no efficient strategy has been proposed. The present pilot study aimed to examine the feasibility and efficiency of an innovative strategy named endoclip papilloplasty to repair the damaged ampulla and recover SO function. The advantage of this device is that it can be rotated clockwise or counterclockwise by turning the handle until the correct position is achieved. Another advantage is if the clip is not in desired position, it may be re-opened and repositioned. Once satisfying clip positioning is achieved, the clip can be firmly attached to the tissue by pulling the slider back until tactile resistance is felt in the handle.

The investigators will recruit patients according to admission criteria and exclusion criteria. The participants underwent SOM before, immediately after EST, and 3 weeks after EST with endoclip papilloplasty. The participants were followed for 3 days during hospitalized. Complications including perforation, bleeding, and PEP were recorded. Blood routine, pancreatic enzymes (amylase and lipase), and liver function (serum alanine aminotransferase, aspartate aminotransferase, r-glutamyl transpeptidase, and alkaline phosphatase) were tested at 4 and 24 h after ERCP. All participants were followed at 3 weeks. Symptoms were examined and blood tests as above were repeated ahead of stents retrieval and sphincter of Oddi monitoring through duodenoscope.

ELIGIBILITY:
Inclusion Criteria:

- 1)18-85 years of age; 2) informed consent obtained before ERCP; 3) CBD diameter ≥12 mm; 4) CBD gallstones visualized at magnetic resonance cholangiopancreatography (MRCP) with at least one gallstone ≥10 mm (transverse diameter)

Exclusion Criteria:

1. gallstone transverse diameter >35 mm, which is not appropriate to be extracted;
2. history of previous sphincterotomy, previous EPBD;
3. accompanied with choledochoduodenal fistula, coagulopathy, anticoagulant/antiplatelet therapy, or Billroth II or Roux-en-Y reconstruction;
4. papilla located deep within a diverticulum;
5. small papilla and short intramural segment, which was not suitable for large EST;
6. medications known to affect the SO (calcium channel blockers, nitrates, opiates, and anticholinergics) taken within 48 h of the procedure;
7. benign or malignant biliary stricture.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a prospective pilot study of consecutive patients with CBD gallstones (transverse diameter ≥10 mm) who were treated at the Gastroenterology Department of Peking University Third Hospital by large-EST combined with endoclip papilloplasty between May 2018 and March 2019.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
SO manometric data | Before operation、During operation、Three weeks after operation
  The comparison of the SO manometric data before and after the procedure

SECONDARY OUTCOMES:
Frequency of use of ML and the incidence of adverse events | Three weeks after operation
  Measure the frequency of use of ML and the incidence of adverse events, and to evaluate the healing of the ampulla.

CONTACTS AND LOCATIONS:
Overall Officials: Yonghui Huang, MD, Study Director — Peking University Third Hosptial
Locations (1):
- Peking University Third Hosptial, Beijing, Beijing Municipality, China